CLINICAL TRIAL: NCT06937268
Title: Exploratory Analysis of DOTATATE PET for Meningioma Radiation Planning
Brief Title: DOTATATE PET for Meningioma Radiation Planning
Acronym: DOTATATE-RT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H22-03733
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Meningioma
MeSH Terms: conditions — Meningioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DOTATATE-PET scan (Experimental)
  Interventions: Diagnostic Test: DOTATATE-PET scan

INTERVENTIONS:
Diagnostic Test: DOTATATE-PET scan — DOTATATE tracer PET scan for meningioma

SUMMARY:
68Ga-DOTATATE-based radionuclides are a novel modality in the diagnosis and treatment of central nervous system meningioma. DOTATATE is a ligand for the SSTR (somatostatin receptor), which is expressed in meningioma but not in normal brain or bone. It is also more effective than MRI in delineating tumor, which is the current imaging standard for assessing meningioma. For radiation planning, it can help to reduce the risk of geometrical miss, identify area that require dose-escalation, and reduce dose to normal tissue. The purpose of the study is to compare the radiation therapy (RT) contouring and planning for meningioma with and without the use of 68Ga-DOTATATE-PET

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Able and willing to comply with the study procedures
* Intact meningioma requiring definitive radiation
* Post-operative meningioma requiring adjuvant radiation
* No prior radiation therapy or medical therapy directed at the tumour

Exclusion Criteria:

* Breastfeeding or pregnancy
* Claustrophobia or inability to lie still in a supine position
* Unwillingness or inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Target radiation volume | 2 years
  The volume of gross total volume (GTV), clinical target volume (CTV), planned target volume (PTV) contours, and volume of dose exposure to normal brain tissue using standard imaging and DOTATE-PET scan

SECONDARY OUTCOMES:
Local control | 2 years
Progression-free survival | 2 years
Perceived usefulness by radiation oncologist | 2 years
Adverse event | 2 years
Rate of DOTATATE-scan completion | 2 years
Extent of post-operative disease volume compared to MRI | 2 years
Overall survival | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- BC Cancer - Vancouver, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided